CLINICAL TRIAL: NCT01332019
Title: A Dose-Frequency Blinded, Multicenter, Extension Study to Determine the Long-Term Safety and Efficacy of PEGylated Interferon Beta-1a (BIIB017) in Subjects With Relapsing Multiple Sclerosis
Brief Title: Long-Term Safety and Efficacy Study of Peginterferon Beta-1a
Acronym: ATTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105MS302; 2010-024477-39 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-04-08 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Subcutaneous; Extension; Interferon; MS; PEGylated; Injectable; SC; PEG; peginterferon beta-1a; Relapsing
MeSH Terms: conditions — Recurrence | interventions — peginterferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peginterferon beta-1a Q4W (Experimental): 125 µg peginterferon beta-1a administered by subcutaneous (SC) injection every 4 weeks (Q4W) for at least 2 years and up to 4 years.
  Interventions: Drug: peginterferon beta-1a
- peginterferon beta-1a Q2W (Experimental): 125 μg peginterferon beta-1a administered by SC injection every 2 weeks (Q2W) for at least 2 years and up to 4 years.
  Interventions: Drug: peginterferon beta-1a

INTERVENTIONS:
Drug: peginterferon beta-1a — Administered as specified in the treatment arm
  Other Names: PEGylated Interferon beta-1a; Plegridy; PEG IFN β-1a; BIIB017

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of peginterferon beta-1a (BIIB017) in participants originally treated in Study 105MS301 (NCT00906399) who continue peginterferon beta-1a treatment. The secondary objective of this study is to describe long-term multiple sclerosis (MS) outcomes in participants originally treated in Study 105MS301 (NCT00906399) who continue peginterferon beta-1a treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have completed the study treatment and visit schedule through Week 96 in Study 105MS301 (NCT00906399).

Key Exclusion Criteria:

* Subjects exceeding more than 6 weeks since completion of the Week 96 visit of Study 105MS301 (NCT00906399).
* Subjects with any clinically significant laboratory abnormalities, malignancies, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease
* Pregnant or nursing women.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2011-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (121):
- United States (7):
  - Research Site, Atlanta, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Franklin, Tennessee
- Research Site, Sint-Truiden, Belgium
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Santiago, Chile
- Colombia (2):
  - Research Site, Barranquilla
  - Research Site, Bogotá
- Research Site, Zagreb, Croatia
- Czechia (7):
  - Research Site, Brno
  - Research Site, Havffov
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Ostrava-Vitkovice
  - Research Site, Prague
  - Research Site, Teplice
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (4):
  - Research Site, Amiens
  - Research Site, Bouches-du-Rhone
  - Research Site, Clermont-Ferrand
  - Research Site, Nice
- Research Site, Tbilisi, Georgia
- Germany (10):
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Erbach im Odenwald
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Marberg
  - Research Site, Prien am Chiemsee
  - Research Site, Ulm
  - Research Site, Westerstede
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- India (15):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Indore, Madhyr Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Amritsar, Punjab
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Mangalore
  - Research Site, Navi Mumbai
  - Research Site, New Delhi
  - Research Site, Saket
- Research Site, Riga, Latvia
- Mexico (5):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Héroes de Padierna
  - Research Site, Mexico City
  - Research Site, Monterrey
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Nieuwegein
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Dunedin
- Peru (2):
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (14):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gmina Końskie
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Plewiska
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Campulung Muscel
  - Research Site, Sibiu
  - Research Site, Târgu Mureş
- Russia (10):
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kransodar
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Smolensk
  - Research Site, Ufa
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
- Spain (4):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Ukraine (10):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Simferopol
  - Research Site, Ternopil
  - Research Site, Vinnytsia
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Sheffield

REFERENCES:
- [Derived] Arnold DL, Shang S, Dong Q, Meergans M, Naylor ML. Peginterferon beta-1a every 2 weeks increased achievement of no evidence of disease activity over 4 years in the ADVANCE and ATTAIN studies in patients with relapsing-remitting multiple sclerosis. Ther Adv Neurol Disord. 2018 Aug 28;11:1756286418795085. doi: 10.1177/1756286418795085. eCollection 2018. PMID 30181780
- [Derived] Seddighzadeh A, Hung S, Selmaj K, Cui Y, Liu S, Sperling B, Calabresi PA. Single-use autoinjector for peginterferon-beta1a treatment of relapsing-remitting multiple sclerosis: safety, tolerability and patient evaluation data from the Phase IIIb ATTAIN study. Expert Opin Drug Deliv. 2014 Nov;11(11):1713-20. doi: 10.1517/17425247.2014.944159. Epub 2014 Jul 29. PMID 25073663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study 105MS302 (NCT01332019) is an extension study and includes participants previously randomized to Study 105MS301 (NCT00906399). Only participants in Study 105MS301 who completed the study treatment and visit schedule through Week 96 were eligible for entry into this study.
Pre-assignment Details: Participants continued BIIB017 at the same dosage regimen they were following during treatment year 2 of Study 105MS301: BIIB017 125 μg subcutaneously (SC) every 2 weeks (Q2W) or every 4 weeks (Q4W). A major change in study design was introduced in Amendment 3 of the protocol, which switched all ongoing subjects dosing Q4W to dosing Q2W.
Groups:
- BIIB017 Q4W: 125 µg BIIB017 administered by SC injection Q4W for at least 2 years and up to 4 years.
- BIIB017 Q2W: 125 µg BIIB017 administered by SC injection Q2W for at least 2 years and up to 4 years.
Period: Overall Study
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Started | 530 | 547
Completed | 417 | 425
Not Completed | 113 | 122
Not completed — Was Not Dosed | 1 | 0
Not completed — Other | 16 | 18
Not completed — Death | 2 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Withdrawal by Subject | 73 | 71
Not completed — Lost to Follow-up | 4 | 7
Not completed — Adverse Event | 13 | 22

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: who entered Study 105MS302 and received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BIIB017 Q4W | BIIB017 Q2W | Total
Number analyzed (Participants) | 529 | 547 | 1076
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.95) | 38.7 (9.59) | 38.4 (9.77)
Age, Customized [Number; unit: participants]
  20-29 years | 131 | 107 | 238
  30-39 years | 165 | 180 | 345
  40-49 years | 150 | 172 | 322
  50-59 years | 80 | 83 | 163
  60-65 years | 3 | 5 | 8
Gender [Count of Participants; unit: Participants]
  Female | 378 | 397 | 775
  Male | 151 | 150 | 301

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Serious AEs, and Discontinuations Due to AEs
Description: AE: any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. SAE: any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, placed the participant at immediate risk of death (a life threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, could have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed in the definition above. Data collected after Amendment 3 took effect were excluded for participants enrolled into study 105MS302 on every 4 week dosing, but not excluded for participants enrolled on every 2 week dosing.
Time Frame: up to 4 years
Population: Safety population: all participants who received at least 1 dose of study drug. For participants who switched to alternative MS medications, data after switch and 14 days after last dose of study treatment are excluded.
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  Any event | 471 | 478
  Moderate or severe event | 343 | 348
  Severe event | 74 | 73
  Event related to study treatment | 400 | 399
  Serious event | 113 | 90
  Discontinuing study treatment due to an event | 18 | 26
  Withdrawing from study due to an event | 14 | 23

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Hematology Laboratory Abnormalities
Description: Data collected after Amendment 3 took effect were excluded for participants enrolled into study 105MS302 on every 4 week dosing, but not excluded for participants enrolled on every 2 week dosing.
Time Frame: up to 4 years
Population: Safety population: all participants who received at least 1 dose of study drug and at least 1 post-baseline value for given parameter.
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 528 | 547
participants
  White blood cells < 3.0*10^9/L | 28 | 86
  White blood cells ≥ 16.0*10^9/L | 13 | 4
  Lymphocytes < 0.8*10^9/L | 41 | 62
  Lymphocytes < 0.5*10^9/L | 2 | 7
  Lymphocytes > 12*10^9/L | 0 | 0
  Segmented neutrophils ≤ 1*10^9/L | 8 | 16
  Segmented neutrophils < 1.5*10^9/L | 31 | 84
  Segmented neutrophils ≥ 12*10^9/L | 18 | 5
  Total absolute neutrophils ≤ 1*10^9/L | 8 | 15
  Total absolute neutrophils < 1.5*10^9/L | 31 | 83
  Total absolute neutrophils ≥ 12*10^9/L | 18 | 5
  Red blood cells ≤ 3.3*10^12/L | 1 | 7
  Red blood cells ≥ 6.8*10^12/L | 0 | 0
  Hemoglobin ≤ 100 g/L | 33 | 35
  Platelet count ≤ 100*10^9/L | 3 | 11
  Platelet count ≥ 600*10^9/L | 2 | 2

3. Primary Outcome: Number of Participants With Shifts From Baseline: Liver Function Laboratory Values
Description: Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high. For participants who switched to alternative MS medications, data after switch and 14 days after last dose of study treatment are excluded. Data collected after Amendment 3 took effect were excluded for participants enrolled into study 105MS302 on every 4 week dosing, but not excluded for participants enrolled on every 2 week dosing. ALT=alanine aminotransferase; AST=aspartate aminotransferase; GGT=gamma-glutamyl transferase.
Time Frame: Baseline (BIIB017 Treatment Baseline from Study 105MS301) up to 4 years
Population: Safety population: all participants who received at least 1 dose of study drug; n=number of participants whose baseline value was not low (or high) and who had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  ALT: shift to low; n=528, 546 | 3 | 3
  ALT: shift to high; n=487, 497 | 119 | 153
  AST: shift to low; n=528, 546 | 10 | 8
  AST: shift to high; n=514, 530 | 75 | 110
  Total bilirubin: shift to low; n=512, 517 | 94 | 76
  Total bilirubin: shift to high; n=511, 535 | 22 | 16
  GGT: shift to low; n=529, 545 | 16 | 6
  GGT: shift to high; n=512, 528 | 73 | 97
  Alkaline phosphatase: shift to low; n=522, 543 | 4 | 5
  Alkaline phosphatase: shift to high; n=516, 536 | 28 | 26
  Lactate dehydrogenase: shift to low; n=529, 547 | 0 | 0
  Lactate dehydrogenase: shift to high; n=524, 541 | 18 | 30

4. Primary Outcome: Number of Participants With Shifts From Baseline: Kidney Function and Other Blood Chemistry
Description: Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high. For participants who switched to alternative MS medications, data after switch and 14 days after last dose of study treatment are excluded. Data collected after Amendment 3 took effect were excluded for participants enrolled into study 105MS302 on every 4 week dosing, but not excluded for participants enrolled on every 2 week dosing. TSH=thyroid stimulating hormone.
Time Frame: Baseline (BIIB017 Treatment Baseline from Study 105MS301) up to 4 years
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  Blood urea nitrogen: shift to low; n=529, 546 | 0 | 1
  Blood urea nitrogen: shift to high; n=527, 543 | 16 | 20
  Creatinine: shift to low; n=529, 547 | 0 | 1
  Creatinine: shift to high; n=528, 545 | 15 | 8
  Bicarbonate: shift to low; n=523, 540 | 49 | 64
  Bicarbonate: shift to high; n=529, 544 | 0 | 0
  Sodium: shift to low; n=529, 546 | 0 | 3
  Sodium: shift to high; n=524, 544 | 39 | 46
  Potassium: shift to low; n=527, 544 | 13 | 21
  Potassium: shift to high; n=528, 546 | 17 | 20
  Chloride: shift to low; n=529, 546 | 1 | 2
  Chloride: shift to high; n=528, 547 | 0 | 3
  Glucose: shift to low; n=522, 539 | 54 | 51
  Glucose: shift to high; n=506, 513 | 304 | 311
  TSH: shift to low; n=515, 533 | 47 | 30
  TSH: shift to high; n=518, 539 | 37 | 55

5. Primary Outcome: Number of Participants With Shifts From Baseline: Urinalysis
Description: Shift to low includes normal to low, high to low, and unknown to low. Shift to high/positive includes normal to high/positive, low to high/positive, negative to high/positive, and unknown to high/positive. For participants who switched to alternative MS medications, data after switch and 14 days after last dose of study treatment are excluded. Data collected after Amendment 3 took effect were excluded for participants enrolled into study 105MS302 on every 4 week dosing, but not excluded for participants enrolled on every 2 week dosing. Pos=positive; RBC=red blood cells; WBC=white blood cells.
Time Frame: Baseline (BIIB017 Treatment Baseline from Study 105MS301) up to 4 years
Population: Safety population: all participants who received at least 1 dose of study drug; n=number of participants whose baseline value was not low or high/positive and who had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  Specific gravity: shift to low; n=525, 545 | 2 | 1
  Specific gravity: shift to high/pos; n=528,547 | 13 | 3
  pH: shift to low; n=529, 547 | 0 | 0
  pH: shift to high/pos; n=528, 547 | 6 | 4
  Color: shift to high/pos; n=516, 529 | 33 | 36
  Blood: shift to high/pos; n=469, 495 | 159 | 167
  Glucose: shift to high/pos; n=521, 542 | 28 | 25
  Ketones: shift to high/pos; n=510, 530 | 64 | 73
  Protein: shift to high/pos; n=380, 391 | 270 | 277
  RBC: shift to high/pos; n=419, 402 | 110 | 106
  WBC: shift to high/pos; n=472, 495 | 116 | 130
  Bilirubin: shift to high/pos; n=529, 547 | 0 | 1
  Nitrite: shift to high/pos; n=508, 519 | 84 | 94
  Urobilinogen: shift to high/pos; n=529, 546 | 7 | 13

6. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the examining neurologist. The annualized relapse rate is calculated as the total number of relapses occurred during the period for all participants, divided by the total number of person-years followed in the period.
Time Frame: up to 4 years
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: relapses per person-years
Units Other Than Participants: Relapses
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
Number analyzed (Relapses) | 232 | 200
relapses per person-years | 0.189 [0.154 to 0.231] | 0.142 [0.114 to 0.177]
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Based on negative binomial regression for each treatment group, with adjustment for EDSS (<4 vs. >=4), relapse rate (based on 1 year before 105MS301 and 105MS301), and age (<40 vs. >=40) at 105MS302 baseline; Test type: Superiority or Other; p = 0.0203, negative binomial regression — q2w/q4w; rate ratio = 0.755, 95% CI 2-sided [0.595 to 0.957]

7. Secondary Outcome: Percentage of Participants Who Relapsed
Description: Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the examining neurologist. New or recurrent neurologic symptoms that occur less than 30 days following the onset of a relapse were considered part of the same relapse. Participants who did not experience a relapse prior to switching to alternative MS medications, withdrew from study, or Amendment 3 (A3) took effect were censored at the time of switch/withdrawal/A3 effective date.
Time Frame: Up to 4 years
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
percentage of participants
  Did not relapse | 71 | 77
  Relapsed | 29 | 23
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; q2w/q4w; Test type: Superiority or Other; p = 0.0201, Cox proportion hazards model — Based on Cox proportion hazards model, adjusted for EDSS (<4 vs >= 4), age (<40 vs >=40), relapse rate (based on one year before 105MS301 and 105MS301), and gadolinium (Gd) enhancing lesions (presence vs. absence) at 105MS302 baseline; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.59 to 0.96]

8. Secondary Outcome: Number of New or Newly Enlarging T2 Hyperintense Lesions
Description: The total number of new or newly enlarging T2 hyperintense lesions (from Study 105MS302 Baseline) as assessed by magnetic resonance imaging (MRI). Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Week 48, Week 96
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment; n=number of participants with an assessment at given timepoint.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 481 | 493
lesions
  Week 48; n=481, 493 | 4.4 (8.19) | 1.9 (4.50)
  Week 96; n=411, 407 | 8.9 (16.64) | 3.9 (9.37)
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 48; Test type: Superiority or Other; p < 0.0001, negative binomial regression — Lesion mean ratio (95% CI) and p-value for comparison between the every 2 weeks group and the every 4 weeks group, based on negative binomial regression, adjusted for 105MS302 baseline number of T2 lesions; lesion mean ratio = 0.51, 95% CI 2-sided [0.41 to 0.63]
Statistical Analysis 2: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 96; Test type: Superiority or Other; p < 0.0001, negative binomial regression — Lesion mean ratio (95% CI) and p-value for comparison between the every 2 weeks group and the every 4 weeks group, based on negative binomial regression, adjusted for 302 baseline number of T2 lesions; lesion mean ratio = 0.49, 95% CI 2-sided [0.39 to 0.62]

9. Secondary Outcome: Number of New Active Lesions
Description: The number of new active lesions as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
lesions
  Week 48; n=481, 493 | 4.4 (8.25) | 2.0 (4.62)
  Week 96; n=411, 406 | 9.0 (16.88) | 3.9 (9.47)
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 48; Test type: Superiority or Other; p < 0.0001, negative binomial regression — Lesion mean ratio (95% CI) and p-value for comparison between the every 2 weeks group and the every 4 weeks group, based on negative binomial regression, adjusted for 105MS302 baseline number of Gd lesions; lesion mean ratio = 0.54, 95% CI 2-sided [0.43 to 0.68]
Statistical Analysis 2: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 96; Test type: Superiority or Other; p < 0.0001, negative binomial regression — [p-value comment as in outcome 9, analysis 1]; lesion mean ratio = 0.55, 95% CI 2-sided [0.43 to 0.71]

10. Secondary Outcome: Number of New T1 Hypointense Lesions
Description: The total number of new T1 hypointense lesions as assessed by MRI.
Time Frame: Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
lesions
  Week 49; n=481, 493 | 1.4 (3.02) | 0.8 (2.18)
  Week 96; n=411, 406 | 2.8 (5.92) | 1.5 (4.14)
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 48; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value for comparison between the every 2 weeks group and the every 4 weeks group, based on multiple logit regression, adjusted for 302 baseline number of T1 lesions
Statistical Analysis 2: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 96; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Number of Gd-Enhancing Lesions
Description: The number of Gd-enhancing lesions as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
lesions
  Baseline; n=528, 543 | 0.6 (1.85) | 0.2 (1.07)
  Week 48; n=481, 493 | 0.7 (2.07) | 0.2 (1.42)
  Week 96; n=411, 407 | 0.8 (2.59) | 0.2 (0.89)
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 48; Test type: Superiority or Other; p = 0.0012, Regression, Logistic — p-value for comparison between the every 2 weeks group and the every 4 weeks group, based on multiple logit regression, adjusted for 302 baseline number of Gd-enhancing lesion
Statistical Analysis 2: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Week 96; Test type: Superiority or Other; p = 0.0026, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Volume of T2 Hyperintense Lesions
Description: The volume of T2 hyperintense lesions as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
cm^3
  Baseline; n=528, 543 | 11.4742 (13.55811) | 9.9678 (11.41807)
  Week 48; n=481, 493 | 11.7421 (13.91774) | 9.8335 (11.05029)
  Week 96; n=411, 407 | 12.0257 (13.91056) | 9.9487 (10.97208)

13. Secondary Outcome: Volume of T1 Hypointense Lesions
Description: The volume of T1 hypointense lesions as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
cm^3
  Baseline; n=528, 543 | 3.9869 (6.29557) | 3.6320 (5.47465)
  Week 48; n=481, 493 | 4.3062 (6.92839) | 3.6529 (5.19027)
  Week 96; n=411, 407 | 4.3171 (6.70107) | 3.7494 (5.21314)

14. Secondary Outcome: Volume of Gd-Enhancing Lesions
Description: The volume of Gd-enhancing lesions as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
cm^3
  Baseline; n=528, 543 | 0.0911 (0.30013) | 0.0348 (0.17344)
  Week 48; n=481, 493 | 0.1172 (0.42762) | 0.0477 (0.31479)
  Week 96; n=411, 407 | 0.1346 (0.50580) | 0.0357 (0.14976)

15. Secondary Outcome: Percentage Change of Whole Brain Volume
Description: Percentage change of whole brain volume as assessed by MRI. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
percentage change
  Change at Week 48; n=402, 418 | -0.522 (0.6205) | -0.453 (0.8127)
  Change at Week 96; n=365, 358 | -0.835 (1.0785) | -0.788 (1.1912)

16. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS)
Description: Change from Baseline in disability as measured by the Expanded Disability Status Scale (EDSS). The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. Data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 12, 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=516, 535 | 2.43 (1.346) | 2.35 (1.299)
  Change at Week 12; n=503, 524 | 0.02 (0.388) | 0.00 (0.450)
  Change at Week 24; n=500, 519 | 0.02 (0.449) | 0.00 (0.486)
  Change at Week 48; n=488, 497 | 0.08 (0.564) | 0.03 (0.510)
  Change at Week 72; n=468, 484 | 0.13 (0.629) | 0.06 (0.484)
  Change at Week 96; n=429, 446 | 0.15 (0.618) | 0.09 (0.563)
  Change at Week 120; n=187, 205 | 0.19 (0.700) | 0.10 (0.538)
  Change at Week 144; n=90, 98 | 0.23 (0.720) | 0.10 (0.587)
  Change at Week 168; n=21, 25 | 0.24 (0.889) | 0.18 (0.454)

17. Secondary Outcome: Time to Sustained Disability Progression
Description: Estimated proportion of participants with progression and time to progression based on the Kaplan-Meier product limit method. Sustained disability progression is defined as: at least a 1.0 point increase on the EDSS from 105MS302 baseline EDSS ≥ 1.0 that is sustained for 24 weeks, or at least a 1.5 point increase on the EDSS from 105MS302 baseline EDSS = 0 that is sustained for 24 weeks. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. Participants were censored at the time of withdrawal/switch/A3 effective date if they withdrew from study, switched to alternative MS medication, or Amendment 3 took effect without a progression.
Time Frame: Weeks 12, 24, 28, 72, 96, 120, 144, 168
Population: Participants in the ITT population (all participants who were assigned a treatment and received at least 1 dose of study treatment) with disability progression.
Measure: Number; unit: proportion of participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 63 | 38
proportion of participants
  Progressed at 12 weeks | 0.023 | 0.007
  Progressed at 24 weeks | 0.046 | 0.023
  Progressed at 48 weeks | 0.079 | 0.045
  Progressed at 72 weeks | 0.103 | 0.057
  Progressed at 96 weeks | 0.115 | 0.069
  Progressed at 120 weeks | 0.147 | 0.085
  Progressed at 144 weeks | 0.161 | 0.096
  Progressed at 168 weeks | NA — Estimated proportion is not calculated if the number of participants at risk is less than 30. | NA — Estimated proportion is not calculated if the number of participants at risk is less than 30.
Statistical Analysis 1: Comparison: BIIB017 Q4W vs BIIB017 Q2W; Test type: Superiority or Other; p = 0.0060, Cox Proportional Hazards model — Based on Cox Proportional Hazards model, adjusted for 105MS302 baseline EDSS and age (<40 vs >=40); Cox Proportional Hazard = 0.57, 95% CI 2-sided [0.38 to 0.85] — q2w/q4w

18. Secondary Outcome: Change From Baseline in Symbol Digit Modalities Test (SDMT)
Description: SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 (worst) to 110 (best).
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment; n=participants with an assessment at given timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=523, 543 | 52.134 (17.7653) | 52.744 (17.6994)
  Change at Week 24; n=508, 530 | -0.313 (8.5862) | -1.106 (8.1292)
  Change at Week 48; n=493, 509 | -0.365 (9.3557) | -0.864 (8.6059)
  Change at Week 72; n=472, 489 | -0.625 (8.8037) | -1.012 (8.5038)
  Change at Week 96; n=435, 450 | -0.340 (8.7817) | -0.231 (9.3148)
  Change at Week 120; n=190, 203 | -1.305 (8.9248) | -1.099 (9.5425)
  Change at Week 144; n=88, 96 | -1.727 (7.7900) | -0.906 (10.8367)
  Change at Week 168; n=21, 25 | -4.000 (10.4403) | -3.840 (13.4712)

19. Secondary Outcome: Change From Baseline in Multiple Sclerosis Impact Scale (MSIS)-29 Physical Score
Description: The 29-item MSIS-29 is a disease-specific participant-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Responses use a 5-point Likert scale ranging from 1 to 5. All questions are to be answered. The physical well being assessment portion of the MSIS-29 consists of 20 questions in which participants rate the impact of MS on their day-to-day life during the past two weeks from 1=no impact to 5=extreme impact for a total score of 20-100. A lower total score indicates less physically-related impact while a higher total score indicates greater physically-related impact on a participant's functioning. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=527, 544 | 20.494 (19.8290) | 20.218 (19.0264)
  Change at Week 24; n=513, 534 | -0.152 (9.3332) | 0.552 (10.0147)
  Change at Week 48; n=498, 510 | 0.462 (10.7054) | 0.545 (10.6342)
  Change at Week 72; n=474, 491 | 0.937 (11.5682) | 0.684 (12.4690)
  Change at Week 96; n=437, 452 | 1.471 (10.8997) | 1.190 (11.4005)
  Change at Week 120; n=193, 205 | 2.654 (14.2983) | 0.116 (10.4382)
  Change at Week 144; n=88, 98 | 0.327 (10.5888) | 0.051 (12.1417)
  Change at Week 168; n=20, 26 | 2.250 (7.3292) | -0.288 (13.5615)

20. Secondary Outcome: Change From Baseline in 12-Item Short Form Health Survey (SF-12) Mental Component Score (MCS)
Description: The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. MCS computed using the scores of 12 questions and range from 0 to 100, where a 0 score indicates the lowest level of health and 100 indicates the highest level of health. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=527, 544 | 47.803 (10.2111) | 48.591 (10.3624)
  Change at Week 24; n=514, 535 | 0.396 (7.5967) | -0.734 (8.3567)
  Change at Week 48; n=498, 510 | 0.409 (8.4442) | -0.690 (8.3903)
  Change at Week 72; n=474, 491 | 0.242 (9.3223) | -0.162 (9.0676)
  Change at Week 96; n=437, 452 | -0.141 (9.4833) | 0.014 (8.8856)
  Change at Week 120; n=193, 205 | -1.223 (10.4664) | 0.616 (7.5313)
  Change at Week 144; n=88, 98 | 0.346 (8.6814) | 0.110 (8.0301)
  Change at Week 168; n=20, 26 | -0.451 (8.8575) | 0.294 (9.7505)

21. Secondary Outcome: Change From Baseline in SF-12 Physical Component Score (PCS)
Description: The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. PCS was computed using the scores of 12 questions and range from 0 to 100, where a 0 score indicates the lowest level of health and 100 indicates the highest level of health. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=527, 544 | 45.154 (9.4474) | 44.902 (9.9312)
  Change at Week 24; n=514, 535 | 0.138 (6.0841) | 0.337 (5.7878)
  Change at Week 48; n=498, 510 | -0.351 (6.1785) | 0.214 (5.8377)
  Change at Week 72; n=474, 491 | -0.270 (6.6319) | -0.169 (6.3824)
  Change at Week 96; n=437, 452 | -0.150 (6.6971) | -0.138 (6.4453)
  Change at Week 120; n=193, 205 | -0.118 (7.8826) | 0.021 (6.1354)
  Change at Week 144; n=88, 98 | -0.256 (5.7252) | 0.118 (6.7830)
  Change at Week 168; n=20, 26 | -1.558 (7.6525) | 0.152 (7.5206)

22. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D) Index Score
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Scores of 1, 2, or 3 are possible responses for each of 5 questions (1=no problems, 2=some problems, 3=severe problems). A scoring formula developed by the EuroQol Group is then used to assign utility values for each participant's Health State Profile. A summary index score (EQ-5D index score) is derived from the 5 questions by conversion with this scoring formula and a table of scores. EQ-5D Summary Index values ranged from -0.6 (worst health state) to 1.00 (perfect health state). Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=527, 544 | 0.76 (0.230) | 0.76 (0.230)
  Change at Week 24; n=514, 534 | 0.00 (0.159) | 0.00 (0.171)
  Change at Week 48; n=498, 510 | -0.01 (0.159) | 0.00 (0.171)
  Change at Week 72; n=472, 491 | -0.01 (0.158) | 0.00 (0.179)
  Change at Week 96; n=436, 452 | -0.01 (0.156) | -0.01 (0.195)
  Change at Week 120; n=193, 205 | -0.02 (0.190) | 0.00 (0.165)
  Change at Week 144; n=88, 98 | 0.00 (0.169) | 0.01 (0.166)
  Change at Week 168; n=21, 26 | 0.00 (0.080) | 0.02 (0.137)

23. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS)
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.' The scale was normalized to a scale of 0 to 1, with higher values indicating a better health state. Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: Baseline (start of 105MS302), Weeks 24, 48, 72, 96, 120, 144, 168
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Baseline; n=527, 542 | 77.07 (17.623) | 77.33 (18.348)
  Change at Week 24; n=511, 532 | -0.22 (11.411) | -0.98 (12.064)
  Change at Week 48; n=498, 508 | -0.81 (12.828) | -0.93 (12.719)
  Change at Week 72; n=472, 490 | -0.59 (12.735) | -1.89 (15.270)
  Change at Week 96; n=436, 450 | -1.10 (14.266) | -2.20 (14.095)
  Change at Week 120; n=193, 204 | -0.47 (12.714) | -0.88 (12.793)
  Change at Week 144; n=88, 97 | -0.31 (14.247) | -0.87 (14.865)
  Change at Week 168; n=21, 26 | 1.38 (14.925) | 0.46 (12.602)

24. Secondary Outcome: Number of Relapses Requiring IV Steroid Use
Description: Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: up to 4 years
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment
Measure: Number; unit: relapses
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
relapses | 217 | 181

25. Secondary Outcome: Number of MS-Related Hospitalizations
Description: Observed data after participants switched to alternative MS medications or after Amendment 3 took effect are excluded.
Time Frame: up to 4 years
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment
Measure: Number; unit: hospitalizations
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
hospitalizations | 113 | 81

26. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: How Tolerable or Intolerable Do You Find the Medication?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "How tolerable or intolerable do you find the medication?" answers were numerically rated from 1 (extremely intolerable) to 10 (extremely tolerable). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 6.8 (2.36) | 7.0 (2.21)
  Year 2; n=425, 430 | 7.2 (2.28) | 7.1 (2.27)
  Year 3; n=82, 88 | 7.5 (2.46) | 7.3 (2.17)

27. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: How Convenient or Inconvenient Is It to Take Your Medication as Instructed?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "How convenient or inconvenient is it to take your medication as instructed?" answers were numerically rated from 1 (extremely inconvenient) to 10 (extremely convenient). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.2 (2.09) | 8.0 (2.12)
  Year 2; n=426, 430 | 8.3 (1.98) | 8.2 (2.05)
  Year 3; n=82, 88 | 8.3 (2.05) | 8.0 (2.08)

28. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: How Convenient or Inconvenient Is It to Take Your Medication Every 2 Weeks?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "How convenient or inconvenient is it to take your medication every 2 weeks?" answers were numerically rated from 1 (extremely inconvenient) to 10 (extremely convenient). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.4 (2.02) | 8.4 (1.99)
  Year 2; n=426, 430 | 8.6 (1.93) | 8.4 (2.06)
  Year 3; n=82, 88 | 8.6 (2.00) | 8.5 (1.79)

29. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: Overall, How Satisfied or Dissatisfied Are You With This Medication?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "Overall, how satisfied or dissatisfied are you with this medication?" answers were numerically rated from 1 (extremely dissatisfied) to 10 (extremely satisfied). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 7.9 (2.04) | 8.1 (1.97)
  Year 2; n=426, 430 | 8.2 (2.04) | 8.3 (2.00)
  Year 3; n=82, 88 | 8.2 (2.00) | 8.6 (1.60)

30. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: How Satisfied or Dissatisfied Are You With the Injection Frequency (Every 2 Weeks)?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "How satisfied or dissatisfied are you with the injection frequency (every 2 weeks)?" answers were numerically rated from 1 (extremely dissatisfied) to 10 (extremely satisfied). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.4 (1.92) | 8.3 (1.98)
  Year 2; n=426, 430 | 8.5 (1.89) | 8.3 (2.07)
  Year 3; n=82, 88 | 8.7 (1.99) | 8.6 (1.59)

31. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: How Likely Would You Be to Continue to Use This Medication?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "How likely would you be to continue to use this medication?" answers were numerically rated from 1 (extremely unlikely) to 10 (extremely likely). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.5 (2.11) | 8.6 (2.00)
  Year 2; n=426, 430 | 8.1 (2.67) | 8.3 (2.58)
  Year 3; n=82, 88 | 8.5 (2.39) | 8.8 (2.00)

32. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: This Medication Enables Me to Focus More on Myself and My Family Rather Than My MS.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "This Medication Enables Me to Focus More on Myself and My Family Rather Than My MS," answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 7.3 (2.52) | 7.8 (2.21)
  Year 2; n=426, 430 | 7.8 (2.35) | 7.8 (2.31)
  Year 3; n=82, 88 | 8.0 (2.44) | 8.3 (2.00)

33. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: This Medication Makes It Easy For Me to Carry Out My Daily Responsibilities.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "This medication makes it easy for me to carry out my daily responsibilities (ie, going to work, doing household chores or caring for my family)," answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 247
units on a scale
  Year 1; n=482, 496 | 7.4 (2.44) | 7.7 (2.33)
  Year 2; n=426, 429 | 7.8 (2.32) | 7.7 (2.35)
  Year 3; n=82, 88 | 7.9 (2.57) | 8.3 (2.07)

34. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: The Twice a Month Dosing Makes It More Convenient for Me to Travel/Vacation.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "The twice a month dosing makes it more convenient for me to travel/vacation," answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.2 (2.21) | 8.2 (2.13)
  Year 2; n=426, 430 | 8.3 (2.20) | 8.2 (2.21)
  Year 3; n=82, 88 | 8.6 (1.97) | 8.5 (1.86)

35. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: The Twice a Month Dosing Enables Me to Be More Spontaneous and Flexible.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "The twice a month dosing enables me to be more spontaneous and flexible," answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.1 (2.20) | 8.2 (2.09)
  Year 2; n=426, 430 | 8.3 (2.12) | 8.2 (2.12)
  Year 3; n=82, 88 | 8.5 (2.17) | 8.4 (1.93)

36. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: This Medication Improves My Self-Confidence and Self-Reliance.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "This medication improves my self-confidence and self-reliance," answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 7.5 (2.47) | 7.7 (2.29)
  Year 2; n=426, 429 | 7.9 (2.50) | 7.9 (2.31)
  Year 3; n=82, 88 | 8.1 (2.45) | 8.4 (1.98)

37. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: I Am Satisfied With the Dosing Frequency of This Medication.
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the statement "I am satisfied with the dosing frequency (2 times per month) of this medication" answers were numerically rated from 1 (strongly disagree) to 10 (strongly agree). Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
units on a scale
  Year 1; n=482, 496 | 8.4 (1.98) | 8.5 (1.94)
  Year 2; n=425, 430 | 8.7 (1.83) | 8.5 (2.06)
  Year 3; n=82, 88 | 8.8 (1.87) | 8.7 (1.81)

38. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: Over the Past 4 Weeks, Did You Miss Any of Your Injections?
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "Over the past 4 weeks, did you miss any of your injections?" answer choices were given as "none missed," "miss 1 injection," or "miss 2 injections." Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  Year 1: none missed; n=482, 493 | 474 | 487
  Year 1: 1 missed; n=482, 493 | 8 | 4
  Year 1: 2 missed; n=482, 493 | 0 | 2
  Year 2: none missed; n=426, 429 | 422 | 426
  Year 2: 1 missed; n=426, 429 | 3 | 2
  Year 2: 2 missed; n=426, 429 | 1 | 1
  Year 3: none missed; n=81, 88 | 79 | 86
  Year 3: 1 missed; n=81, 88 | 0 | 1
  Year 3: 2 missed; n=81, 88 | 2 | 1

39. Secondary Outcome: Summary of Participant-Reported Treatment Satisfaction: Main Reason for Missed Injections
Description: Participants completed a Treatment Satisfaction Questionnaire composed of a range of 14 questions regarding the participant's perception of treatment satisfaction at the end of each year of treatment. For the question "Main reason for missed injections?" answer choices were given as "medication side effects," "injection pain," "forget to take medication," "tired of taking injections," "don't think medication is working," or "other." Data after Amendment 3 took effect are excluded.
Time Frame: Year 1, Year 2, Year 3
Population: ITT population: all participants who were assigned a treatment and received at least 1 dose of study treatment; n=participants with an assessment who missed at least 1 injection at given timepoint.
Measure: Number; unit: participants
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Number analyzed (Participants) | 529 | 547
participants
  Year 1: medication side effects; n=8, 6 | 0 | 1
  Year 1: injection pain; n=8, 6 | 0 | 0
  Year 1: forget to take medication; n=8, 6 | 2 | 1
  Year 1: tired of taking injections; n=8, 6 | 0 | 0
  Year 1: don't think medication is working; n=8, 6 | 0 | 0
  Year 1: other; n=8, 6 | 6 | 4
  Year 2: medication side effects; n=4, 3 | 1 | 1
  Year 2: injection pain; n=4, 3 | 0 | 0
  Year 2: forget to take medication; n=4, 3 | 1 | 1
  Year 2: tired of taking injections; n=4, 3 | 0 | 0
  Year 2: don't think medication is working; n=4, 3 | 0 | 0
  Year 2: other; n=4, 3 | 2 | 1
  Year 3: medication side effects; n=2, 2 | 0 | 0
  Year 3: injection pain; n=2, 2 | 0 | 0
  Year 3: forget to take medication; n=2, 2 | 0 | 0
  Year 3: tired of taking injections; n=2, 2 | 1 | 1
  Year 3: don't think medication is working; n=2, 2 | 0 | 0
  Year 3: other; n=2, 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 4 years
Description: All treatment-emergent events are presented. (An event was considered to be treatment emergent if it had an onset date on or after the date of first study treatment or if it was present prior to start of study treatment and subsequently worsened.)
Arm/Group | BIIB017 Q4W | BIIB017 Q2W
Serious Adverse Events (participants affected / at risk) | 114/529 | 91/547
Other Adverse Events (participants affected / at risk) | 435/529 | 438/547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB017 Q4W (N=529) | BIIB017 Q2W (N=547)
Angina pectoris (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Heterophoria (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Infectious thyroiditis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 3
Facial neuralgia (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 2
Multiple sclerosis relapse (Nervous system disorders) | 83 | 57
Secondary progressive multiple sclerosis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Status epilepticus (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Uhthoff's phenomenon (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bipolar 1 disorder (Psychiatric disorders) | 1 | 0
Catatonia (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB017 Q4W (N=529) | BIIB017 Q2W (N=547)
Nausea (Gastrointestinal disorders) | 25 | 34
Asthenia (General disorders) | 64 | 45
Chills (General disorders) | 70 | 58
Fatigue (General disorders) | 40 | 52
Influenza like illness (General disorders) | 234 | 234
Injection site erythema (General disorders) | 222 | 224
Injection site pain (General disorders) | 38 | 34
Injection site pruritus (General disorders) | 24 | 34
Pyrexia (General disorders) | 147 | 132
Nasopharyngitis (Infections and infestations) | 68 | 49
Upper respiratory tract infection (Infections and infestations) | 18 | 34
Urinary tract infection (Infections and infestations) | 51 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 52
Back pain (Musculoskeletal and connective tissue disorders) | 53 | 57
Myalgia (Musculoskeletal and connective tissue disorders) | 65 | 67
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 | 55
Headache (Nervous system disorders) | 152 | 161
Hypoaesthesia (Nervous system disorders) | 31 | 28
Multiple sclerosis relapse (Nervous system disorders) | 155 | 130
Paraesthesia (Nervous system disorders) | 31 | 20
Depression (Psychiatric disorders) | 27 | 26
Insomnia (Psychiatric disorders) | 27 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.